CLINICAL TRIAL: NCT00193505
Title: Phase II Trial of Ifosfamide/Carboplatin/Etoposide/Rituxan Followed by Zevalin in the Treatment of Patients With Relapsed/Refractory Intermediate Grade B-Cell Lymphoma
Brief Title: Ifosfamide/Carboplatin/Etoposide/Rituxan Followed by Zevalin in Relapsed/Refractory Intermediate Grade B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Biogen (Industry)
Responsible Party: John Hainsworth, MD, Sarah Cannon Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LYM 27; 106-P092
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Non-Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Ifosfamide; Carboplatin; Etoposide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ifosfamide
Drug: Carboplatin
Drug: Etoposide
Drug: Rituximab
Drug: 90Y Zevalin

SUMMARY:
In this Multicenter trial, we will evaluate the feasibility, toxicity, and efficacy of treatment with 90Y Zevalin following a short course of salvage chemotherapy in patients with relapsed/refractory intermediate grade B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

* Ifosfamide + Carboplatin + Etoposide + Rituximab

Patients showing no response to this combination regimen will receive 90Y Zevalin after two cycles or when progression is clearly documented. In responding patients, four cycles will be administered, followed by 90Y Zevalin.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Intermediate grade CD20-positive B-cell non-Hodgkin's lymphoma
* Persistent lymphoma after one or two previous chemotherapy regimens
* Patients should not be considered candidates for high-dose chemotherapy
* Ability to perform activities of daily living with assistance
* Measurable or evaluable disease
* Age > 18 years
* Adequate bone marrow, liver and kidney function

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Patients with impaired bone marrow reserve
* Female patients who are pregnant or lactating
* Serious active infection at the time of treatment
* Any other serious underlying condition
* Brain or meningeal) with lymphoma
* HIV or AIDS-related lymphoma
* Received external beam radiation therapy to > 25% of active bone marrow.
* History of other cancers, either active or treated

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
complete response rate

SECONDARY OUTCOMES:
progression-free survival
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States